CLINICAL TRIAL: NCT05356078
Title: Association Between Prescription of Antidepressants and Delirium in the Elderly : Analysis From the World Health Organization Global Database
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco20220103
Record Dates: First submitted 2022-01-31; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Antidepressive Agents; Aged; Delirium
MeSH Terms: conditions — Delirium | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antidepressant — "Delirium" event reported in the World Health Organization global database in subjects aged over 65 years taking antidepressants, comparative analysis by antidepressant class

SUMMARY:
Delirium is a frequent reason for hospitalisation of the elderly. Associations between the prescription of some medicines and the risk of delirium have already been demonstrated.

Antidepressants are widely prescribed in the elderly because of the frequency of anxiety-depressive symptoms in this population, where there are high pharmacokinetic and pharmacodynamic variability.

However, the association between antidepressants and the risk of delirium remains poorly understood.

Based on the analysis from the World Health Organization global database, the main objective of this study is to investigate the association between the different classes of antidepressants and the occurrence of the " delirium " event reported in the database.

A disproportionality analysis will be performed. It will aim to assess whether some classes of antidepressants, and within these classes some molecules, are associated with a greater risk of delirium.

ELIGIBILITY:
Inclusion Criteria:

* be over 65 years old
* taking antidepressants
* to have presented delirium

Exclusion Criteria:

-

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and over who presented with delirium on antidepressants
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-06-03 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of the studied population | 03/01/2022
  From the WORLD HEALTH ORGANIZATION Vigibase pharmacovigilance database, the investigators select all patients over 65 years old.
  Then among them, the investigators report :
  * Antidepressants use by class (Non-selective monoamine reuptake inhibitors, Selective serotonin reuptake inhibitors, Selective serotonin-norepinephrine reuptake Inhibitors, Alpha-2-adrenergic receptor antagonists, Monoamine oxidase inhibitors, other antidepressants)
  * Delirium event
  * Co-prescription (Opioids, Antipsychotics, Anxiolytics, Hynotics)
  * Comorbidities (Constipation, acute retention of urine, hyponatraemia etc...)
Analysis of the association between antidepressant classes and delirium reporting, among subjects aged 65 or older | 03/01/2022
  A disproportionality analysis is carried out in multivariate analysis, taking into account a certain number of confounding factors (co-prescriptions and comorbidities)

SECONDARY OUTCOMES:
Analysis by age group | 03/01/2022
  Investigators study the association between antidepressant classes and delirium reporting for the age group 65-74 and for the age group 75 and over.
  A disproportionality analysis is carried out in multivariate analysis, taking into account a certain number of confounding factors (co-prescriptions and comorbidities)
Analysis of the co-reporting of delirium and hyponatraemia | 03/01/2022
  Investigators study the association between antidepressant classes and co-reporting of delirium and hyponatraemia among subjects aged 65 or older.
  A disproportionality analysis is carried out in multivariate analysis, taking into account a certain number of confounding factors (co-prescriptions and comorbidities).
Analysis of the most prescribed antidepressant | 03/01/2022
  Investigators study the association between most prescribed antidepressants and delirium reporting among patients aged 65 or older.
  We identified most prescribed antidepressants as those with more than 1000 cases reported in VigiBase®.
  A disproportionality analysis is carried out in multivariate analysis, taking into account a certain number of confounding factors (co-prescriptions and comorbidities).

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No